CLINICAL TRIAL: NCT02086721
Title: Phase I Clinical Study Combining L19-IL2 With Stereotactic Ablative Body Radiotherapy in Patients With Oligometastatic Solid Tumor.
Brief Title: Phase I Clinical Study Combining L19-IL2 With SABR in Patients With Oligometastatic Solid Tumor
Acronym: L19-IL2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L19-IL2
Record Dates: First submitted 2013-09-03; First posted 2014-03-13 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Solid Tumour
MeSH Terms: interventions — L19-IL2 immunocytokine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oligometastatic cancer patients; N=18 (Experimental)
  Interventions: Drug: L19-IL2

INTERVENTIONS:
Drug: L19-IL2 — Patients receive a schedule of 1 x 30 Gy, 3 x 15-20 Gy; 5 x 12 Gy; 8 x 7.5 Gy; to the 80 % or 100 % isodose.
  Step -1: Toxicity of 10 Mio IU of L19-IL2 (n=3-6)10 Mio IU of L19-IL2 (max. 6 cycles) via i.v. bolus injection.
  Toxicity scored at every i.v. drug administration and on day 7, 14 and 21. Step 1: Toxicity of 15 Mio IU of L19-IL2 (n=3-6)(max. 6 cycles) via i.v. bolus injection.
  Step 2: Toxicity of 22.5 Mio IU of L19-IL2 (n=3-6)(max. 6 cycles) via i.v. bolus injection.
  Toxicity scored at every i.v. drug administration and on day 7, 14 and 21 of the cycle.
  Step 3: Expansion cohort of the maximally tolerable dose (n=10) Administration of the maximally tolerable dose of L19-IL2(max. 6 cycles) via i.v. bolus injection.
  Toxicity scored at every i.v. drug administration and on day 7, 14 and 21 of the cycle.

SUMMARY:
The formation of metastasis is responsible for as much as 90% of cancer-associated mortality. In spite of recent advances in oncologic therapy, approximately 50 % of the lung cancer patients have already overt disseminated cancer at diagnosis. Additionally, numerous patients with locoregional disease initially treated with curative intent develop (oligo)metastases during the course of disease. In both instances, these stage IV patients are generally considered to be incurable and mostly treated palliatively.

Oligometastases, defined as 1-5 sites of active disease on whole body imaging, was coined to refer to isolated sites of metastasis resembling limited tumor metastatic capacity. The implication of this concept is that local cancer treatments are curative in a proportion of patients with metastases and that incorporating local therapy is a conceptually attractive approach. In several, but not all, academic centers the standard treatment of patients with oligometastases in good general health is standard chemotherapy followed by surgery or by Stereotactic Ablative Body Radiotherapy (SABR) with radical dose on the macroscopic visible tumors.

The widespread introduction of SABR and of minimally invasive surgery has fuelled research in treating patients with oligometastases. Indeed, local control of metastases can be obtained in virtually all parts of the body with a low proportion of patients experiencing severe side effects. In the few prospective studies published to date, approximately 20% of patients remained free of recurrence several years after treatment when all sites of disease were targeted by radiation.

Along with standard anti-cancer therapeutic modalities like chemotherapy and radiotherapy (RT), immunotherapy has recently gained a lot of attention.

Angiogenesis is one of the hallmarks of cancer, and therefore, considerable efforts have been made to exploit this unique target for selective drug delivery. One of the appealing targets for both approaches is the splice variant of fibronectin containing extra domain B (EDB), which is abundantly expressed in vascular endothelial cells of a variety of primary tumors as well as metastases , but virtually absent in normal tissues. Recently, a human recombinant scFv fragment directed against EDB, designated L19, was developed and subsequently combined with the pro-inflammatory interleukin-2 (IL2), resulting in the immunocytokine L19-IL2. L19-IL2 delivers high doses of IL2 to the (metastatic) tumor site(s) exploiting the selective expression of EDB on newly formed blood vessels. Interleukin-2 (IL2) plays an essential role in the activation phases of both specific and natural immune responses. Even though it has no direct cytotoxic effects on cancer cells, it can induce tumor regression by stimulating a potent cell-mediated response. In summary, L19-IL2 is an immunocytokine which will stimulate immune response specifically in tumors with angiogenesis and tissue remodeling.

Radiotherapy is a particularly interesting partner for immunotherapy, since it can be harnessed to specifically modify the immunogenicity of the primary tumors and their microenvironment, in the attempt to generate an in situ immunization of the host against a patient's own cancer. Our hypothesis is that three independent therapeutic approaches will synergize to improve dramatically survival in patients with oligometastases of solid tumors.

DETAILED DESCRIPTION:
1. Tumor vasculature Profound differences exist between vascular endothelium and surrounding stroma of normal tissues and tumors. Tumor vasculature is extremely disorganized and tortuous. Vascular shunts are frequent, and distinguishing arterioles from venules can be challenging. Apart from the architecture, the blood flow itself is strikingly altered: it can be sluggish, sometimes stationary or even reverse. The endothelium in tumors proliferates rapidly and contributes to active angiogenesis. The direct contact of the tumor endothelium with the host's blood pool makes this site a unique target for selective drug delivery.
2. L19 Fibronectin (FN) is a broadly present soluble constituent of plasma and other body fluids. FN usually exists as a dimer formed by two nearly identical (approximately 250 kDa) subunits covalently linked near their C-terminus by a pair of disulfide bonds. Even though FN molecules are the product of a single gene, the resulting protein can exist in multiple forms that arise from alternative spicing of pre-mRNA that can generate up to 20 variants in humans. Splicing occurs in 3 regions of the FN gene, leading to inclusion or exclusion of either one of the two type III repeats, named EDB and EDA. The 91 amino acid sequence of EDB is identical in mice, rats, rabbits, dogs and humans. EDB-containing FN is dispensable during embryogenesis, but is thought to play a modulating role in the growth of connective tissues. In adults, EDB-FN is highly expressed in normal tissues during angiogenesis, but not in mature vessels. Furthermore, EDB-containing FN is abundantly found in solid tumors. It is mainly produced by tumor cells and deposited in the subendothelial extracellular matrix of solid tumors and hematological malignancies.

   L19 is the single chain (scFv) human antibody that specifically targets EDB-FN. Antibody fragments in small scFv formats are useful and versatile tools with various advantages including rapid blood clearance and easy manipulation for antibody engineering. The L19 antibody has been shown to recognize and target EDB-FN in vivo both in animal models and patients. In past years, the L19 antibody has been conjugated with numerous agents, including therapeutic radionuclides, and cytokines.
3. Interleukin-2 Cytokines are a heterogeneous group of soluble small polypeptides or glycoproteins exerting pleiotropic or redundant effects promoting growth, differentiation, and activation of normal cells. Cytokines produced by immune cells may have pro- or anti-inflammatory and immune-modulatory activities. In malignant diseases, cytokine production and release can be affected by the tumor itself and/or therapeutic interventions. Cytokines may also display potent anticancer activities, but are frequently hampered by treatment-related toxicities prohibiting dose-escalation to therapeutically effective concentrations.

   Interleukin-2 (IL2) plays an essential role in the activation phases of both specific and natural immune responses. Even though it has no direct cytotoxic effects on cancer cells, it can induce tumor regression by stimulating a potent cell-mediated response. As such, IL2 is one of the treatment options in metastatic renal cell carcinoma patients.
4. L19-IL2 In order to overcome toxicity while simultaneously delivering therapeutic doses of IL2 to the tumor issue, the elegant option of combining the anti-EDB scFv L19 antibody with IL2 was pursued. It has been shown that the L19-IL2 conjugate mediates the selective delivery and accumulation of IL2 at tumor endothelial cells, where the EDB antigen is expressed during angiogenesis, leading to a dramatic increase of the therapeutic efficacy of IL2. In the first preclinical study, 80% of the xenograft tumors (including teratocarcinoma and small cell lung cancer) tackled with L19-IL2 were subsequently composed of connective and necrotic tissue. At the same time an increase in the levels of interferon-gamma and of cytotoxic lymphocytes, macrophages and natural killer cells was found. These histological and therapeutic effects were underlined in a orthotopic pancreatic cancer model treated with the antibody-cytokine conjugate. One year later, this response percentage was repeated in Ramos lymphoma xenografts treated with L19-IL2 and the anti-CD20 antibody rituximab whereby a complete remission lasting for more than one year was found in 4 of the 5 mice treated.

In a recent phase I/II clinical trial, the use of L19-IL2 was proven safe in a variety of stage IV malignancies with a recommended dose of 22.5 Mio IU. Furthermore, it was safely combined with dacarbazine in stage IV melanoma patients maintaining the same recommended dose level. In the first study, the overall objective response rate was reported to be 51% after two cycles, and in the second this rate was 28% with one complete response still ongoing 21 months after treatment initiation.

At present, three phase I/II clinical trials on L19-IL2 alone or in combination with chemotherapy for patients with metastatic melanoma (ClinicalTrials.gov numbers: NCT01055522 and NCT01253096) and pancreatic cancer (ClinicalTrials.gov number: NCT01198522) are ongoing.

Summary Study Design

Details on SABR:

Prescribed dose is risk adapted to the metastatic localization and closeness to organs at risk (in accordance with local protocol of MAASTRO clinic). Patients will receive a dose schedule of 1 x 30 Gy, 3 x 15-20 Gy; 5 x 12 Gy; 8 x 7.5 Gy; to the 80 % or 100 % isodose which should encompass the periphery of the PTV as closely as possible. Maximum dose is not restricted but volumes with a dose higher than 105% must be located within the gross tumor. The minimum dose allowed is EQD2α/ẞ10 =60 Gy, an ablative dose with EQD2iso=≥ 87.5Gy10 should always be the objective. Treatment will be delivered with intensity modulated arcs treatments.

Step -1: Assessment of the toxicity of 10 Mio IU of L19-IL2 (n=3-6); this step is only chosen when dose-limiting toxicity occurs in Step 1.

Administration of 10 Mio IU of L19-IL2 given on day 1, 3 and 5 of each 21-day cycle (max. 6 cycles) via i.v. bolus injection starting within one week after completion of SABR.

Toxicity will be scored at every intravenous (i.v.) drug administration and on day 7, 14 and 21 of the cycle, according to the CTCAE4.0 scoring system. Hematology, liver and kidney function will be controlled on day 1, 3, and 5 prior to L19-IL2 administration, and on day 7, 14 and 21.

When in 0/3 patients a toxicity of grade 2 or more has occurred step 1 is considered safe. If in 1/3 or more patients a grade 2 or more toxicity has occurred, 3 more patients will be included in this step. If another grade 2 or more toxicity occurs in 1/3 or more patients, the study will be stopped. When at maximum 1/6 patients experience grade 2 toxicity, this step will be considered safe. When step 1 is considered safe, step 2 will be initiated.

Step 1: Assessment of the toxicity of 15 Mio IU of L19-IL2 (n=3-6) Administration of 15 Mio IU of L19-IL2 given on day 1, 3 and 5 of each 21-day cycle (max. 6 cycles) via i.v. bolus injection starting within one week after completion of SABR.

Toxicity will be scored at every i.v. drug administration and on day 7, 14 and 21 of the cycle, according to the CTCAE4.0 scoring system. Hematology, liver and kidney function will be controlled on day 1, 3, and 5 prior to L19-IL2 administration, and on day 7, 14 and 21.

When in 0/3 patients a toxicity of grade 2 or more has occurred step 1 is considered safe. If in 1/3 or more patients a grade 2 or more toxicity has occurred, 3 more patients will be included in this step. If another grade 2 or more toxicity occurs in 1/3 or more patients, the study will be stopped. When at maximum 1/6 patients experience grade 2 toxicity, this step will be considered safe. When step 1 is considered safe, step 2 will be initiated.

Step 2: Assessment of the toxicity of 22.5 Mio IU of L19-IL2 (n=3-6) Administration of 22.5 Mio IU of L19-IL2 given on day 1, 3 and 5 of each 21-day cycle (max. 6 cycles) via i.v. bolus injection starting within one week after completion of SABR.

Toxicity will be scored at every i.v. drug administration and on day 7, 14 and 21 of the cycle, according to the CTCAE4.0 scoring system. Hematology, liver and kidney function will be controlled on day 1, 3, and 5 prior to L19-IL2 administration, and on day 7, 14 and 21.

When in 0/3 patients a toxicity of grade 2 or more has occurred step 1 is considered safe. If in 1/3 or more patients a grade 2 or more toxicity has occurred, 3 more patients will be included in this step. If another grade 2 or more toxicity occurs in 1/3 or more patients, the study will be stopped. When at maximum 1/6 patients experience grade 2 toxicity, this step will be considered safe. When step 1 is considered safe, step 2 will be initiated.

Step 3: Expansion cohort of the maximally tolerable dose (n=10) Administration of the maximally tolerable dose of L19-IL2 given on day 1, 3 and 5 of each 21-day cycle (max. 6 cycles) via i.v. bolus injection starting within one week after completion of SABR.

Toxicity will be scored at every i.v. drug administration and on day 7, 14 and 21 of the cycle, according to the CTCAE4.0 scoring system. Hematology, liver and kidney function will be controlled on day 1, 3, and 5 prior to L19-IL2 administration, and on day 7, 14 and 21.

ELIGIBILITY:
Inclusion criteria:

* Histological or cytological confirmed oligometastatic originating from NSCLC, HNSCC, CRC, RCC and melanoma occurring synchronous (at time of diagnosis) or metachronous (> 6 months after radical treatment for primary tumor; i.e., surgically. A biopsy could be omitted in selected cases if a biopsy is medically contraindicated or unfeasable (e.g. fear of ent-metastasis, lesion not accessible). In this case the diagnosis of metastatic disease should be certified using an alternative approach (e.g. imaging..)
* determination of possible activating mutations (e.g., ALK/EGFR/ROS in NSCLC, and BRAF, NRAS and KIT in melanoma);
* All oligometastatic tumor sites (including brain) are eligible;
* ≤ 5 metastases, or 4 if the primary tumor is to be treated concomitantly;
* ≤ 3 metastatic lesions confined to one organ;
* ≤ 2 organ systems affected with metastases;
* WHO performance status 0-2;
* Adequate bone marrow: Normal white blood cell count and formula, normal platelet count, no anemia requiring blood transfusion or erythropoietin;
* Adequate hepatic function: total bilirubin ≤ 1.5 x upper limit of normal (ULN) for the institution; ALT, AST, and alkaline phosphatase ≤ 2.5 x ULN for the institution);
* Adequate renal function: calculated creatinine clearance at least 60 ml/min;
* The patient is capable of complying with study procedures;
* Signed and dated written informed consent;
* Life expectancy of at least 12 weeks;
* For women of childbearing potential, a negative pregnancy test prior to the first dose of study treatment;
* Men and women with reproductive potential must be willing to practice acceptable methods of birth control during the study and for up to 12 weeks after the last dose of study medication.

Exclusion criteria

* Other oligometastatic (hormone-sensitive) solid tumors;
* Previous radiotherapy to an area that would be re-treated by SABR;
* Previous systemic treatment to treat recurrent disease;
* Other active malignancy or malignancy within the last 2 years (with exception of localized skin basal/squamous cell carcinoma, bladder in situ carcinoma);
* History of allergy to intravenously administered proteins/peptides/antibodies;
* HIV infection, active infection, or active hepatitis;
* Chronic use of corticosteroids used in the management of cancer or non-cancer-related illness;
* Acute or sub-acute coronary syndromes within the last year, accute inflammatory heart disease, heart insufficiency or irreversible cardiac arrhythmias;
* Impaired cardiac function defined as left ventricular ejection fraction (LVEF) <50% (or below the study site's lower limit of normal) as measured by MUGA of ECHO. (LVEF measurements dating back up to 8 weeks will be acceptable in the absence of intercurrent use of potentially cardiotoxic treatment of cardiac medical history
* Uncontrolled hypertensive disease
* History or evidence of active autoimmune disease;
* Severe diabetic retinopathy (38);
* Major trauma including surgery within 4 weeks prior to entering the study;
* Any underlying medical or psychiatric condition which in the opinion of the investigator will make administration of study drug hazardous or hinder the interpretation of study results (e.g., AE);
* Unstable or serious concurrent uncontrolled medical conditions;
* Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Toxicity (CTCAE 4.0) | three months

SECONDARY OUTCOMES:
Progression-Free survival | 3 months
Local control rate | 3 months
non-invasive response evaluation using PET | 3 months
Quality of life | 3 months
Correlation of outcome measures with PET-imaging | 3 months
correlation of outcome measures with immunological markers in tumor tissue. | 3 months
Overall survival | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, MD, PhD., Principal Investigator — MAASTR clinic
Locations (1):
- MAASTRO clinic, Maastricht, Limburg, Netherlands